CLINICAL TRIAL: NCT05323838
Title: Influence of Co-diagnosis of Chronic Fatigue Syndrome in Patients With Fibromyalgia on Physical Activity, Quality of Life and Immunoneuroendocrine Response.
Brief Title: Influence of Co-diagnosis of Chronic Fatigue Syndrome in Patients With Fibromyalgia.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Eduardo Otero Calderón, Staff Scientist, Research, University of Extremadura
Other Study IDs: TesisEDUFM
Record Dates: First submitted 2022-03-18; First posted 2022-04-12 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic | interventions — Accelerometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Healthy Women: Aged-matched control group of healthy women.
  Interventions: Behavioral: Subjective quality of live; Procedure: Blood extraction; Behavioral: Accelerometry
- Only Fibromyalgia: Patients diagnosed only with fibromyalgia.
  Interventions: Behavioral: Subjective quality of live; Procedure: Blood extraction; Behavioral: Accelerometry; Dietary Supplement: Synbiotic complement
- Fibromyalgia and Chronic Fatigue Syndrome: Patients diagnosed with fibromyalgia and chronic fatigue syndrome.
  Interventions: Behavioral: Subjective quality of live; Procedure: Blood extraction; Behavioral: Accelerometry; Dietary Supplement: Synbiotic complement

INTERVENTIONS:
Behavioral: Subjective quality of live — The groups fill out scientifically validated questionnaires to know the differences in perceived stress, anxiety, quality of life, depression, quality of sleep, pain, fatigue, and impact of the disease on daily life.
Procedure: Blood extraction — Blood collection by qualified personnel.
Behavioral: Accelerometry — To know the objective differences between physical activity/sedentary lifestyle, caloric expenditure and quality of sleep, we used the accelerometry technique
Dietary Supplement: Synbiotic complement — On two separate days, the "baseline-tests" and "final-tests" were conducted. All participants performed a series of tests, before which they had to fast. The order and schedule (8 am) of the tests was the same for the "final-test" and the same materials and procedures were used. A period of 30 consecutive days elapsed between the base-line and final tests, during which the participants had to ingest their supplement (synbiotic).
  Groups: Fibromyalgia and Chronic Fatigue Syndrome; Only Fibromyalgia

SUMMARY:
The purpose of this study is to evaluate differences in neuroimmunoendocrine response and quality of live in patients diagnosed with Fibromyalgia, with or without a co-diagnosis of Chronic Fatigue Syndrome.

DETAILED DESCRIPTION:
The limited literature published in concordant relation affects the chronic fatigue syndrome comorbidity in the daily life of fibromyalgia patients leads us to design this study with the main objective of evaluating differences in the quality of life associated with pain and stress, mainly in relation to levels of physical activity, sedentary lifestyle and sleep in patients diagnosed with fibromyalgia, with or without a parallel co-diagnosis of chronic fatigue syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia and/or Chronic Fatigue Syndrome diagnosis by rheumatologists or internal medicine professionals.
* Age not less than 40 years old and not more than 65 years old.

Exclusion Criteria:

* Suffering from diagnosed "major depression".
* Suffer diagnosed multiple chemical sensitivity.
* Corticosteroid treatment or anti-cytokine therapies.
* Periodically carry out programmed therapeutic physical activity in the two months prior to the accelerometry tests.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The present investigation is carried out in two experimental groups: patients diagnosed with Fibromyalgia and patients diagnosed with Fibromyalgia and a co-diagnosis of Chronic Fatigue Syndrome, all of them volunteers facilitated through the Fibromyalgia Associations of Badajoz and Cáceres, Extremadura, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2024-11-16 (Estimated)

PRIMARY OUTCOMES:
Differences in perceived anxiety using the State-Trait Anxiety Inventory (STAI) | During the intervention, at day 1.
  State-Trait Anxiety Inventory (STAI) is a self-reported, scientifically validated questionnaire that measures perceived anxiety. The STAI has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Differences in perceived stress using The Perceived Stress Scale (PSS) | During the intervention, at day 1.
  The Perceived Stress Scale (PSS) is a self-reported, scientifically validated questionnaire that measures perceived stress. This scale is a self- report instrument that evaluates the level of perceived stress during the last month, and consists of 14 items with a 5-point response scale (0 = never, 1 = almost never, 2 = once in a while, 3 = often, 4 = very often). The total score of the PSS is obtained by reversing the scores of items 4, 5, 6, 7, 9, 10, and 13 (in the following manner: 0 = 4, 1 = 3, 2 = 2, 3 = 1, and 4 = 0) and subsequently adding the 14 item scores. A higher score indicates a higher level of perceived stress.
Differences in perceived depression using the Beck's Depression Inventory (BDI) | During the intervention, at day 1.
  Beck's Depression Inventory (BDI) is a self-reported, scientifically validated questionnaire that measures perceived depression. Each of the 21 items on the BDI measures the presence and severity of a symptom of depression by requiring a self-rating from 0 to 3. Mild (low) scores are less than 4; moderate (medium) is between 14 and 20, and severe 21 and above. Unless otherwise indicated, the use of "mild," "moderate," and "severe" levels of depression throughout the remainder of this chapter will refer to the aforementioned ranges.
Differences in perceived pain using the Brief Pain Inventory (BPI) | During the intervention, at day 1.
  Brief Pain Inventory (BPI) is a self-reported, scientifically validated questionnaire that measures perceived pain. The BPI starts with a screening question, asking about the presence of pain and a body chart is used to indicate painful regions as well as the worst region. These items aren´t evaluated. This is followed by the core BPI items: the rating scales for pain severity and interference. Numerical rating scales from 0 to 10 are used for all items. The anchors for pain severity scales are 0 = 'no pain' and 10 = 'pain as bad as you can imagine', whilst the interference anchors are 0 = 'no interference' and 10 = 'interferes completely'.
Differences in perceived pain using the Brief Fatigue Inventory (BFI) | During the intervention, at day 1.
  The Brief Fatigue Inventory (BFI) has nine items, with the items measured on 0-10 numeric rating scales. Three items ask patients to rate the severity of their fatigue at its "worst," "usual," and"now" during normal waking hours, with 0 being "no fatigue" and 10 being "fatigue as bad as you can imagine." Six items assess the amount that fatigue has interfered with different aspects of the patient's life during the past 24 hours. The interference items include general activity, mood, walking ability, normal work, relations with other people, and enjoyment of life. The interference items are measured on a 0 -10 scale, with 0 beings "does not interfere" and 10 being "completely interferes."
Differences in subjective quality of sleep using The Pittsburgh Sleep Quality Index (PSQI) | During the intervention, at day 1.
  The Pittsburgh Sleep Quality lndex (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring.
  The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21 " indicating severe difficulties in all areas.
Differences in subjective quality of life using The Healthy Lifestyle and Personal Control Questionnaire (HLPCQ) | During the intervention, at day 1.
  The Healthy Lifestyle and Personal Control Questionnaire (HLPCQ) This is a 26-item tool in which the respondent is asked to indicate the frequency of adopting 26 positively stated lifestyle habits using a Likert-type scale (1=Never or rarely, 2=Sometimes, 3=Often, and 4 = Always).
Differences in perceived anxiety related to Coronavirus Disease (COVID-19) using the Coronavirus Anxiety Scale (CAS) | During the intervention, at day 1.
  The Coronavirus Anxiety Scale is a brief mental health screener that can be used to identify cases of dysfunctional anxiety related to COVID-19. The items measure physiologically-based symptoms that are aroused with coronavirus-related information and thoughts using a 5-point time anchored scale (0=not at all to 4=nearly every day over the last 2 weeks).
Differences in fear of Coronavirus Disease (COVID-19) using the Fear COVID-19 Scale (FCV-19S) | During the intervention, at day 1.
  The Fear of COVID-19 Scale (FCV-19S) is used to identify and intervene early, psychologically, in people with high values of fear of COVID-19. This one-dimensional scale is made up of seven items with a 5-point Likert response ranging from 1 (strongly disagree) to 5 (strongly agree) and the total tables can range between 7 and 35 points. The higher the score, the greater the fear of COVID-19 infection.
Objective differences in physical activity, sedentary lifestyle and sleep using the accelerometer technique (ActiGraph) | Up to 1 week
  An accelerometer is a small device, like a wristwatch, used to measure physical activity level, patterns of activity, sedentary levels, sleep patterns, and the expenditure of calories consumed, basal and total Metabolic Equivalent of Task (METs) used as an assessment of the metabolism of the person wearing it.
Determination of immuno-neuroendocrine parameters (cytokines, catecholamines, and stress hormones) | Through study completion, an average of 2 year
  Cytokines (IL-8, IL-10), catecholamines (such as epinephrine, and norepinephrine) as well as stress hormones (serotonin and cortisol), were analyzed by competitive inhibition enzyme immunoassays (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler GK, Geenen R. Hypothalamic-pituitary-adrenal and autonomic nervous system functioning in fibromyalgia. Rheum Dis Clin North Am. 2005 Feb;31(1):187-202, xi. doi: 10.1016/j.rdc.2004.10.002. PMID 15639063
- [Background] Guillen-Riquelme A, Buela-Casal G. [Meta-analysis of group comparison and meta-analysis of reliability generalization of the State-Trait Anxiety Inventory Questionnaire (STAI)]. Rev Esp Salud Publica. 2014 Jan-Feb;88(1):101-12. doi: 10.4321/S1135-57272014000100007. Spanish. PMID 24728394
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Poquet N, Lin C. The Brief Pain Inventory (BPI). J Physiother. 2016 Jan;62(1):52. doi: 10.1016/j.jphys.2015.07.001. Epub 2015 Aug 21. No abstract available. PMID 26303366
- [Background] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Darviri C, Alexopoulos EC, Artemiadis AK, Tigani X, Kraniotou C, Darvyri P, Chrousos GP. The Healthy Lifestyle and Personal Control Questionnaire (HLPCQ): a novel tool for assessing self-empowerment through a constellation of daily activities. BMC Public Health. 2014 Sep 24;14:995. doi: 10.1186/1471-2458-14-995. PMID 25253039
- [Background] Freedson P, Bowles HR, Troiano R, Haskell W. Assessment of physical activity using wearable monitors: recommendations for monitor calibration and use in the field. Med Sci Sports Exerc. 2012 Jan;44(1 Suppl 1):S1-4. doi: 10.1249/MSS.0b013e3182399b7e. PMID 22157769
- [Background] Lee SA. Coronavirus Anxiety Scale: A brief mental health screener for COVID-19 related anxiety. Death Stud. 2020;44(7):393-401. doi: 10.1080/07481187.2020.1748481. Epub 2020 Apr 16. PMID 32299304
- [Background] Ahorsu DK, Lin CY, Imani V, Saffari M, Griffiths MD, Pakpour AH. The Fear of COVID-19 Scale: Development and Initial Validation. Int J Ment Health Addict. 2022;20(3):1537-1545. doi: 10.1007/s11469-020-00270-8. Epub 2020 Mar 27. PMID 32226353